CLINICAL TRIAL: NCT01541280
Title: Pre-emptive Azacitidine and Donor Lymphocyte Infusions Following Allogeneic Hematopoietic Stem Cell Transplantation for High Risk Acute Myeloid Leukemia and Myelodysplastic Syndrome
Brief Title: VIDAZA-DLI Pre-emptive Azacitidine and Donor Lymphocyte Infusions Following Allogeneic Hematopoietic Stem Cell Transplantation for High Risk Acute Myeloid Leukemia and Myelodysplastic Syndrome
Acronym: VIDAZA-DLI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD 10/07-H
Record Dates: First submitted 2011-12-13; First posted 2012-02-29 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Allogreffe, LAM , MDS; Azacitidine (VidazaÒ); Injection de lymphocytes de donneur (DLI)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Azacitidine (AZA) is to be administered every 28 days beginning day +56 to 100 posttransplant for one year provided the patients has a platelet count of >15 x 109/L without transfusion for at least 2 successive days, and an absolute neutrophil count of >1 x 109/L without growth factor for at least 2 successive days, and no acute GVHD greater than grade I and no clinical evidence of life-threatening infection. AZA is given 32 mg /m²/day subcutaneously for 5 days every 28 days (
Other: DLI — Donor lymphocyte infusion (DLI) is to be given from day +126 (week 18) in patients without immunosuppressive therapy for at least one month and following 3 cycles of AZA, and without clinical signs of GVHD, and without uncontrolled infection and without a recent history of >grade 2 acute GVHD. DLI are schedules every 8 weeks. There are 3 DLI scheduled.
  If first cycle of AZA is postponed beyond day 56 (maximum to Day 100), all subsequent cycles and DLI will be post poned too.

SUMMARY:
Patients included in the study with high risk acute myeloid leukemia or myelodysplastic syndrome as defined will receive an allogeneic transplantation conditioned by either myeloablative or reduced regimen. Following allogeneic transplantation, patients will receive a maintenance regimen combining chemotherapy with azacitidine (aza) and immunotherapy with donor lymphocyte infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high risk acute myeloid leukemia undergoing allogeneic transplantation with either a familial or an unrelated donor.

High risk AML is defined as :

* AML in CR1 with unfavorable cytogenetics defined by complex caryotype, autosomal monosomy combined or not with other cytogenetics abnormalities inv(3)/t(3,3), t(6;9), t(6;11), t(11;19), del(5q), del(7q).
* AML in CR2 or greater remission prior allogeneic transplantation
* AML in PR or relapse prior allogeneic transplantation
* Or Patients with high risk myelodysplastic syndrome undergoing allogeneic transplantation with either a familial or an unrelated donor.

High risk MDS is defined as :

* MDS with intermediate-2 group and higher risk group according to IPSS criteria
* Age 18 - 70 years.
* Availability of an HLA identical family donor or unrelated donor with matching in 10/10 alleles (HLA-A, B, C, DRB1, DQB1) or maximum of 1 allele or antigen mismatch OR family donor with maximum 1 allele mismatch.
* Conditioning regimen to allogeneic transplantation may be either myeloablative or reduced.
* Be able to understand and sign informed consent.
* Affiliation number to National Health Care System
* Men and women of childbearing potential must use effective contraception during and up to 3 months after treatment.

Exclusion Criteria:

* The presence of any one exclusion criteria renders the patient ineligible:
* Patient in full relapse post-transplant (>20% blasts in the bone marrow) following allogeneic transplant
* Documented leukemic infiltration of CNS/cerebrospinal fluid.
* Karnofsky performance score below 60%.
* Acute and chronic heart failure (NYHA Class III or IV) or symptomatic ischemic heart disease.

following allogeneic transplant

* Severe liver failure (bilirubin >30 μmoles/L, SGPT > 4 X upper limit of normal).
* Hepatic malignancy in advanced stage.
* Severe neurological or psychiatric disorders
* Acute GVHD grade II-III. Patient with grade I GVHD may be included (see annex 1 for GHVD grade definition).
* Active uncontrolled infection.
* Denied informed consent.
* Treatment with other investigational drugs following allogeneic transplantation.
* No effective contraception
* Lactating females
* Pregnant woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the cumulative incidence of relapse rate | 2 years
  An A'Hern procedure will be used (cf. 11.1): If the number of patients not relapsed at two year will be 18 or more out of 24 patients, the null hypothesis will be rejected and the relapse rate will be considered acceptable.

SECONDARY OUTCOMES:
Evaluation of disease-free survival (DFS) at 2 years from transplantation | 2 years
  Kaplan-Meier method
Measure the overall survival rate at 2 years | 2 years
  Kaplan-Meier method
Cumulative incidence death from leukemia, and non relapse mortality (NRM) | 2 years
  cumulative incidence function for disease free survival at 2 years from transplantation, GVHD, death from leukaemia and non-relapse mortality will be estimated (patients are at risk not only for relapse but can also be "removed" from possible relapse because of competing events such as death in remission (due to infection or GVHD)).
Feasibility and safety of administrating maintenance azacitidine following allogenic transplantaton | 2 years
  To evaluate toxicity induced by the azacitidine and DLI, different parameters will be studied:Cell Blood Count with differential, liver function tests, serum creatinine, BUN and total protein will be performed weekly from the time of initiation of azacitidine administration until completion of the last DLI. Performance Status,Acute GVHD,Bone marrow aspiration with evaluation of morphological response as well as chimerism from peripheral blood will be performed prior starting azacitidine, following 3 cycles of azacitidine and after the seventh cycle and twelfth cycle of azacitidine.
Feasibility and safety of performing prophylactic donor lymphocytes infusion | 2 years
  The relatedness of observed toxicity to DLI will be evaluated and documented:
  * Maximum toxicity with respect to mucositis, liver, kidney, lung, heart, neurological system according to CTC criteria (cf. appendices).
  * Infections (bacteremia, fungemia, invasive fungal infection, CMV reactivation and disease, other viral reactivation or infection).
  * Grade of acute and chronic GVHD (cf. appendices); GVHD is classified according to clinical symptoms, irrespective to the time interval to DLI.
  * Bone marrow aspiration, as well as chimerism in PB.
Incidence and severity of acute and chronic graft-versus-host disease | 2 years
  Symptoms related to GVHD should be reported within the GVHD section of the case reporting files. AE and SAE are documented in the patient's chart
  * on a daily basis, as long as the patient is on ward, and
  * on a weekly to two-monthly basis during outpatient follow up, depending on the frequency of outpatient visits on the respective patient.

CONTACTS AND LOCATIONS:
Overall Officials: Milpied Noel, Professor, Principal Investigator — University Hospital, Bordeaux; Guillaume Thierry, Doctor, Principal Investigator — Nantes University Hospital; Yakoub-Agha Ibrahim, Professor, Principal Investigator — CHU Lille; Huynh Anne, Doctor, Principal Investigator — University Hospital, Toulouse; Blaise Didier, Professor, Principal Investigator — Institut Paoli Calmettes, Marseille; Mohamad Mothy, Professor, Principal Investigator — Hôpital Saint Antoine
Locations (1):
- University Hospital of Nantes, Nantes, France